CLINICAL TRIAL: NCT02441218
Title: Effects of Ivabradine on Cardiovascular Events in Patients With Moderate to Severe Chronic Heart Failure and Left Ventricular Systolic Dysfunction. A Three-year International Multicentre Study
Acronym: SHIFT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL3-16257-063; 2006-000708-18 (EudraCT Number)
Record Dates: First submitted 2015-05-05; First posted 2015-05-12 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Chronic Heart Failure
MeSH Terms: interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ivabradine (Experimental)
  Interventions: Drug: Ivabradine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivabradine — 2.5mg, 5mg or 7.5mg tablets to be taken orally twice daily, at 12-hours intervals, in the morning and in the evening during meals up to 42 months.
  Arms: Ivabradine
Drug: Placebo — Matching placebo tablets to be taken orally twice daily, at 12-hours intervals, in the morning and in the evening during meals up to 42 months.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to demonstrate the superiority of ivabradine over placebo in the reduction of cardiovascular mortality or hospitalisation for worsening heart failure in patients with moderate to severe symptoms of chronic heart failure, a reduced left ventricular ejection fraction and currently receiving recommended therapy for this disease.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Chronic heart failure (NYHA II, III or IV)
* Left ventricular systolic dysfunction (LVEF ≤ 35%)
* Sinus rhythm and resting heart rate ≥ 70 bpm
* Optimal and unchanged CHF medications or dosages

Exclusion Criteria:

* Unstable condition within previous 4 weeks
* Myocardial infarction or coronary revascularisation within previous 2 months
* Stroke or transient cerebral ischaemia within previous 4 weeks
* Congenital heart disease
* Severe valvular disease
* Active myocarditis
* Permanent atrial fibrillation or flutter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6505 (Actual)
Dates: Start 2006-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Hôpital Pitié-Salpétrière, Paris, France
- Göteborg University, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com

REFERENCES:
- [Result] Swedberg K, Komajda M, Bohm M, Borer JS, Ford I, Dubost-Brama A, Lerebours G, Tavazzi L; SHIFT Investigators. Ivabradine and outcomes in chronic heart failure (SHIFT): a randomised placebo-controlled study. Lancet. 2010 Sep 11;376(9744):875-85. doi: 10.1016/S0140-6736(10)61198-1. PMID 20801500
- [Result] Bohm M, Swedberg K, Komajda M, Borer JS, Ford I, Dubost-Brama A, Lerebours G, Tavazzi L; SHIFT Investigators. Heart rate as a risk factor in chronic heart failure (SHIFT): the association between heart rate and outcomes in a randomised placebo-controlled trial. Lancet. 2010 Sep 11;376(9744):886-94. doi: 10.1016/S0140-6736(10)61259-7. PMID 20801495
- [Derived] Tyl B, Lopez Sendon J, Borer JS, Lopez De Sa E, Lerebours G, Varin C, De Montigny A, Pannaux M, Komajda M. Comparison of Outcome Adjudication by Investigators and by a Central End Point Committee in Heart Failure Trials: Experience of the SHIFT Heart Failure Study. Circ Heart Fail. 2020 Jul;13(7):e006720. doi: 10.1161/CIRCHEARTFAILURE.119.006720. Epub 2020 Jun 25. PMID 32580655
- [Derived] Griffiths A, Paracha N, Davies A, Branscombe N, Cowie MR, Sculpher M. Analyzing Health-Related Quality of Life Data to Estimate Parameters for Cost-Effectiveness Models: An Example Using Longitudinal EQ-5D Data from the SHIFT Randomized Controlled Trial. Adv Ther. 2017 Mar;34(3):753-764. doi: 10.1007/s12325-016-0471-x. Epub 2017 Feb 15. PMID 28205056

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The target population was adult patients with stable, moderate to severe chronic heart failure (CHF) and left ventricular systolic dysfunction, with optimal and unchanged CHF medications and dosages for ≥ 4 weeks.
Pre-assignment Details: Following a run-in period of two weeks during which no study treatment was dispensed, the participants were randomised to receive ivabradine or placebo in addition to their usual cardiovascular treatment in double-blind treatment period.
Period: Overall Study
Arm/Group | Ivabradine | Placebo
Started | 3241 | 3264
Completed | 2663 | 2652
Not Completed | 578 | 612
Not completed — Death | 503 | 553
Not completed — Withdrawal by Subject | 73 | 58
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivabradine | Placebo | Total
Number analyzed (Participants) | 3241 | 3264 | 6505
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (11.2) | 60.1 (11.5) | 60.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 779 | 756 | 1535
  Male | 2462 | 2508 | 4970
Beta-blocker intake at randomization [Number; unit: participants]
  Yes | 2897 | 2923 | 5820
  No | 344 | 341 | 685

OUTCOME MEASURES:

1. Primary Outcome: Primary Composite Endpoint: First Event Among Cardiovascular Death (Including Death of Unknown Cause) or Hospitalization for Worsening Heart Failure.
Description: Number of patients having experienced the Primary Composite Endpoint.
Time Frame: All over the study (up to 42 months).
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 3241 | 3264
participants | 793 | 937
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.75 to 0.90] — Estimate of the hazard ratio between treatment groups based on an adjusted Cox proportional hazards model with beta-blocker intake at randomisation as a covariate. P-value: Wald test

2. Secondary Outcome: Cardiovascular Death
Description: Component of the primary composite endpoint
Time Frame: From the date of randomization until the date of death, up to 42 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 3241 | 3264
participants | 449 | 491
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.128, Regression, Cox; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.80 to 1.03] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Hospitalisation for Worsening Heart Failure
Time Frame: From the date of randomization to the date of first documented hospitalisation, up to 42 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 3241 | 3264
participants | 514 | 672
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.66 to 0.83] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: All-cause Mortality
Time Frame: From the date of randomisation to death, up to 42 months.
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 3241 | 3264
participants | 503 | 552
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.092, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.80 to 1.02] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Death From Heart Failure
Description: Component of cardiovascular death
Time Frame: From the date of randomisation to death, up to 42 months.
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 3241 | 3264
participants | 113 | 151
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.0140, Regression, Cox; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.58 to 0.94] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Hospitalisation for Any Cause
Time Frame: From the date of randomisation to the date of first documented hospitalisation, up to 42 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 3241 | 3264
participants | 1231 | 1356
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.0027, Regression, Cox; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.82 to 0.96] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Hospitalisation for Cardiovascular Reason
Time Frame: From the date of randomisation to the first documented hospitalisation, up to 42 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 3241 | 3264
participants | 977 | 1122
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.0002, Regression, Cox; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.78 to 0.92] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Unplanned Hospitalisation for Any Cause
Time Frame: From the date of randomisation to the first documented hospitalisation, up to 42 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 3241 | 3264
participants | 1137 | 1264
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.0013, Regression, Cox; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.81 to 0.95] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Unplanned Hospitalisation for CV Reason
Time Frame: From the date of randomisation to the first documented hospitalisation, up to 42 months.
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 3241 | 3264
participants | 909 | 1047
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p = 0.0002, Regression, Cox; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.77 to 0.92] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Secondary Composite Endpoint
Description: CV death, hospitalisation for worsening HF or hospitalisation for non-fatal myocardial infarction
Time Frame: From the date of randomisation to the date of the first event, up to 42 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Placebo
Number analyzed (Participants) | 3241 | 3264
participants | 825 | 979
Statistical Analysis 1: Comparison: Ivabradine vs Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.74 to 0.89] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From randomisation to death, up to 42 months
Description: The Randomised Set consisted of 6505 patients (3241 patients in the ivabradine group and 3264 patients in the placebo group). The Safety Set consisted of 6492 patients: 13 randomised patients were excluded from the Safety Set because they did not take any study drug (9 patients in the ivabradine group and 4 patients in the placebo group).
Arm/Group | Ivabradine | Placebo
Serious Adverse Events (participants affected / at risk) | 1369/3232 | 1481/3260
Other Adverse Events (participants affected / at risk) | 2062/3232 | 2020/3260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivabradine (N=3232) | Placebo (N=3260)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 8 (8)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Spleen disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 9 (11) | 14 (14)
Acute myocardial infarction (Cardiac disorders) | 62 (65) | 54 (61)
Adams-Stokes syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 51 (61) | 55 (60)
Angina unstable (Cardiac disorders) | 113 (140) | 119 (139)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 126 (139) | 106 (114)
Atrial flutter (Cardiac disorders) | 22 (22) | 19 (20)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 9 (9) | 2 (2)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 7 (7) | 4 (4)
Atrioventricular block third degree (Cardiac disorders) | 8 (8) | 2 (2)
Bradycardia (Cardiac disorders) | 15 (15) | 2 (2)
Cardiac aneurysm (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 506 (766) | 665 (1093)
Cardiac failure acute (Cardiac disorders) | 12 (13) | 5 (5)
Cardiac failure congestive (Cardiac disorders) | 17 (21) | 19 (21)
Cardio-respiratory distress (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 15 (15) | 16 (16)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cor pulmonale (Cardiac disorders) | 1 (4) | 0 (0)
Coronary artery disease (Cardiac disorders) | 5 (5) | 5 (5)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 3 (3)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 2 (2) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 3 (3) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 3 (3)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 57 (63) | 51 (51)
Myocardial ischaemia (Cardiac disorders) | 2 (3) | 3 (3)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1)
Rhythm idioventricular (Cardiac disorders) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 5 (5) | 0 (0)
Sinoatrial block (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 2 (2) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 4 (4) | 5 (5)
Torsade de pointes (Cardiac disorders) | 2 (2) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 3 (3) | 5 (5)
Ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 15 (15) | 9 (9)
Ventricular fibrillation (Cardiac disorders) | 20 (21) | 11 (11)
Ventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 31 (34) | 46 (52)
Gastrointestinal angiodysplasia haemorrhagic (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 3 (3)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 2 (2)
Hyperparathyroidism primary (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 1 (1)
Cataract (Eye disorders) | 9 (11) | 7 (7)
Cataract cortical (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 3 (4) | 1 (1)
Iridocyclitis (Eye disorders) | 0 (0) | 1 (1)
Lens dislocation (Eye disorders) | 1 (1) | 0 (0)
Open angle glaucoma (Eye disorders) | 0 (0) | 1 (1)
Presbyopia (Eye disorders) | 0 (0) | 1 (1)
Retinal artery embolism (Eye disorders) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 1 (1)
Retinopathy proliferative (Eye disorders) | 0 (0) | 1 (1)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colonic haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 5 (5)
Disbacteriosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum duodenal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 4 (4) | 2 (2)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Femoral hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 3 (3) | 3 (3)
Gastric ulcer perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 4 (4) | 4 (4)
Gastritis atrophic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastritis haemorrhagic (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroduodenitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal erosion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 5 (5)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 8 (8) | 8 (9)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 3 (3)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Megacolon (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 5 (5) | 5 (5)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 5 (5)
Polyp colorectal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sigmoiditis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 2 (2)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 (1) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Accidental death (General disorders) | 0 (0) | 1 (1)
Cardiac death (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 5 (5) | 4 (7)
Death (General disorders) | 4 (4) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1)
Implant site inflammation (General disorders) | 1 (1) | 0 (0)
Implant site ulcer (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 5 (5) | 2 (4)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Sudden cardiac death (General disorders) | 73 (73) | 68 (68)
Sudden death (General disorders) | 111 (111) | 119 (119)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 2 (2)
Biliary colic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 7 (7) | 11 (11)
Cholecystitis acute (Hepatobiliary disorders) | 5 (5) | 9 (9)
Cholelithiasis (Hepatobiliary disorders) | 6 (6) | 5 (5)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cytolytic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 3 (3) | 3 (3)
Hepatic congestion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatorenal failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Post cholecystectomy syndrome (Hepatobiliary disorders) | 0 (0) | 2 (2)
Allergic oedema (Immune system disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Cryoglobulinaemia (Immune system disorders) | 0 (0) | 1 (1)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 2 (2)
Ascites infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchiectasis (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 3 (3) | 5 (5)
Bronchitis acute (Infections and infestations) | 10 (11) | 18 (20)
Bronchitis acute viral (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis chronic (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 7 (8) | 7 (8)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
Candida sepsis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 5 (5) | 6 (6)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 1 (1) | 4 (4)
Diabetic gangrene (Infections and infestations) | 5 (5) | 5 (6)
Diverticulitis (Infections and infestations) | 0 (0) | 4 (5)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 2 (2) | 0 (0)
Epidemic nephropathy (Infections and infestations) | 0 (0) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 5 (5) | 7 (8)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 4 (4) | 5 (5)
Gastroenteritis enteroviral (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Graft infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 3 (3)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 4 (4) | 4 (4)
Lower respiratory tract infection (Infections and infestations) | 2 (3) | 4 (4)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 4 (5) | 5 (6)
Lung infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Malaria (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 1 (1)
Obstructive chronic bronchitis with acute exacerbation (Infections and infestations) | 2 (2) | 2 (4)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 3 (4) | 3 (3)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0)
Perianal abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritoneal tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 70 (79) | 65 (69)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia primary atypical (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (3) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 2 (2)
Pulmonary tuberculosis (Infections and infestations) | 3 (3) | 1 (1)
Purulent synovitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 3 (3) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 3 (3)
Pyelonephritis chronic (Infections and infestations) | 4 (4) | 1 (1)
Pyonephrosis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 7 (7) | 7 (8)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 1 (1)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 5 (5)
Septic shock (Infections and infestations) | 1 (1) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 3 (3) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 2 (2)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (4) | 5 (5)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 3 (3)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Closed head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device dislocation (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Diaphragmatic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 7 (8) | 4 (5)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral disc injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple drug overdose accidental (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pacemaker complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Polytraumatism (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Postoperative hernia (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Renal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skeletal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Stent occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Urinary bladder rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound evisceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 0 (0) | 1 (1)
Arteriogram (Investigations) | 2 (2) | 0 (0)
Arteriogram coronary (Investigations) | 24 (24) | 12 (13)
Blood chloride decreased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Carcinoembryonic antigen increased (Investigations) | 0 (0) | 1 (1)
Cardiac electrophysiologic study (Investigations) | 0 (0) | 3 (3)
Cardiac pacemaker evaluation (Investigations) | 1 (1) | 1 (1)
Cardiovascular evaluation (Investigations) | 27 (32) | 27 (31)
Catheterisation cardiac (Investigations) | 0 (0) | 5 (6)
Coagulation time prolonged (Investigations) | 0 (0) | 1 (1)
Colonoscopy (Investigations) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 3 (3) | 0 (0)
Hysteroscopy (Investigations) | 1 (1) | 0 (0)
Investigation (Investigations) | 1 (1) | 2 (2)
Nephrological examination (Investigations) | 1 (1) | 1 (1)
Pregnancy test positive (Investigations) | 0 (0) | 1 (1)
Sleep study (Investigations) | 1 (1) | 1 (1)
Transplant evaluation (Investigations) | 2 (2) | 5 (5)
Ultrasound Doppler (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 23 (25) | 33 (34)
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Diabetic foot (Metabolism and nutrition disorders) | 3 (8) | 8 (8)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Dactylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Chronic lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear cell carcinoma of the kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Malignant mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Oropharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Brain stem haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 5 (5) | 4 (4)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral arteriosclerosis (Nervous system disorders) | 2 (2) | 3 (3)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 3 (3)
Cerebral infarction (Nervous system disorders) | 7 (7) | 12 (13)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 14 (14) | 16 (17)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 2 (2) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Embolic stroke (Nervous system disorders) | 1 (1) | 3 (3)
Encephalitis (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Facial palsy (Nervous system disorders) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 2 (2) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 34 (37) | 46 (48)
Lacunar infarction (Nervous system disorders) | 1 (1) | 3 (3)
Loss of consciousness (Nervous system disorders) | 1 (1) | 4 (4)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 12 (12) | 20 (21)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 0 (0)
Tarsal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 11 (12) | 12 (12)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 3 (3) | 3 (4)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 3 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 1 (1)
Disturbance in social behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Schizophreniform disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 2 (2) | 0 (0)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 1 (2)
Glomerulonephritis chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 14 (14) | 14 (14)
Renal failure acute (Renal and urinary disorders) | 11 (13) | 7 (7)
Renal failure chronic (Renal and urinary disorders) | 2 (2) | 4 (4)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Stress incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (2)
Urinary retention (Renal and urinary disorders) | 1 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 5 (5) | 2 (2)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Phimosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 20 (25) | 25 (31)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (12)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial hyperactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 35 (53) | 33 (50)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Haemopneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 23 (24)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dry gangrene (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Social stay hospitalisation (Social circumstances) | 0 (0) | 1 (1)
Alcohol detoxification (Surgical and medical procedures) | 1 (1) | 0 (0)
Arrhythmia prophylaxis (Surgical and medical procedures) | 1 (1) | 0 (0)
Arterial bypass operation (Surgical and medical procedures) | 1 (1) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac aneurysm repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 4 (4) | 0 (0)
Cardiac rehabilitation therapy (Surgical and medical procedures) | 7 (9) | 7 (10)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 20 (21) | 29 (30)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 1 (2) | 2 (2)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary angioplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1) | 5 (5)
Coronary artery surgery (Surgical and medical procedures) | 12 (12) | 5 (5)
Coronary revascularisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Diabetes mellitus management (Surgical and medical procedures) | 1 (1) | 1 (1)
Ear operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Eventration procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastric banding (Surgical and medical procedures) | 1 (1) | 0 (0)
Heart transplant (Surgical and medical procedures) | 1 (1) | 4 (4)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Implantable defibrillator insertion (Surgical and medical procedures) | 17 (17) | 21 (21)
Implantable defibrillator replacement (Surgical and medical procedures) | 0 (0) | 4 (4)
Incisional hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 2 (2)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 2 (2)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Mitral valve replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Obesity surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Percutaneous coronary intervention (Surgical and medical procedures) | 5 (5) | 2 (2)
Physiotherapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Rehabilitation therapy (Surgical and medical procedures) | 2 (2) | 2 (2)
Renal tumour excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 2 (2) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Ureteral stent removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Weight loss diet (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 3 (4)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 3 (3) | 4 (4)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis obliterans (Vascular disorders) | 3 (3) | 3 (4)
Bleeding varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Blood pressure inadequately controlled (Vascular disorders) | 17 (19) | 13 (13)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 7 (7)
Diabetic macroangiopathy (Vascular disorders) | 0 (0) | 1 (1)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1)
Femoral artery aneurysm (Vascular disorders) | 1 (3) | 0 (0)
Femoral artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 2 (2) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 5 (5) | 5 (5)
Hypertensive emergency (Vascular disorders) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 5 (5)
Iliac artery embolism (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 4 (4) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 15 (15) | 15 (18)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Peripheral embolism (Vascular disorders) | 3 (4) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 5 (7)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivabradine (N=3232) | Placebo (N=3260)
Anaemia (Blood and lymphatic system disorders) | 91 (93) | 92 (96)
Angina pectoris (Cardiac disorders) | 85 (97) | 93 (109)
Atrial fibrillation (Cardiac disorders) | 161 (176) | 123 (138)
Atrioventricular block first degree (Cardiac disorders) | 35 (38) | 36 (42)
Bradycardia (Cardiac disorders) | 134 (142) | 26 (30)
Cardiac failure (Cardiac disorders) | 289 (337) | 299 (369)
Sinus tachycardia (Cardiac disorders) | 40 (45) | 102 (115)
Supraventricular extrasystoles (Cardiac disorders) | 39 (41) | 49 (50)
Ventricular extrasystoles (Cardiac disorders) | 129 (140) | 131 (137)
Ventricular tachycardia (Cardiac disorders) | 34 (37) | 26 (28)
Phosphenes (Eye disorders) | 89 (95) | 16 (18)
Gastritis (Gastrointestinal disorders) | 34 (34) | 36 (36)
Bronchitis (Infections and infestations) | 38 (44) | 34 (40)
Bronchitis acute (Infections and infestations) | 59 (64) | 68 (79)
Influenza (Infections and infestations) | 66 (74) | 68 (76)
Nasopharyngitis (Infections and infestations) | 66 (70) | 70 (85)
Pneumonia (Infections and infestations) | 56 (60) | 69 (78)
Respiratory tract infection (Infections and infestations) | 39 (40) | 25 (28)
Respiratory tract infection viral (Infections and infestations) | 30 (33) | 34 (36)
Upper respiratory tract infection (Infections and infestations) | 33 (35) | 52 (55)
Urinary tract infection (Infections and infestations) | 24 (24) | 37 (40)
Fall (Injury, poisoning and procedural complications) | 36 (40) | 42 (47)
Blood creatinine increased (Investigations) | 55 (58) | 47 (49)
Heart rate decreased (Investigations) | 178 (193) | 45 (46)
Transaminases increased (Investigations) | 46 (48) | 42 (42)
Diabetes mellitus (Metabolism and nutrition disorders) | 32 (32) | 35 (35)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 116 (125) | 115 (125)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 33 (33) | 34 (34)
Hyperkalaemia (Metabolism and nutrition disorders) | 27 (29) | 53 (56)
Hyperuricaemia (Metabolism and nutrition disorders) | 47 (47) | 52 (52)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 24 (24) | 40 (42)
Dizziness (Nervous system disorders) | 55 (62) | 45 (50)
Headache (Nervous system disorders) | 43 (45) | 58 (67)
Renal failure (Renal and urinary disorders) | 50 (53) | 69 (71)
Renal failure chronic (Renal and urinary disorders) | 27 (28) | 45 (45)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 37 (42) | 55 (68)
Cough (Respiratory, thoracic and mediastinal disorders) | 42 (44) | 44 (44)
Blood pressure inadequately controlled (Vascular disorders) | 216 (259) | 188 (215)
Hypotension (Vascular disorders) | 59 (62) | 82 (91)

LIMITATIONS AND CAVEATS:
The section Other Adverse Events (Not including serious) has been completed by the sponsor to include only the Non Serious Adverse Events emergent on treatment during the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review publication and/or communication related to the study results and can require changes. In case of a patent application, the sponsor can delay its authorization for publication or communication of the study results until the date of international registration of the patent.